CLINICAL TRIAL: NCT00501540
Title: A Phase II Clinical and Biological Study of Lithium Carbonate in Patients With Low-Grade Neuroendocrine Tumors
Brief Title: Lithium for Low-Grade Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO07203; R21CA117117-01A2 (NIH); H-2007-0065 (Other: Institutional Review Board); NCI-2011-00616 (Registry Identifier: NCI Trial ID); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison)
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Results first posted 2017-05-03 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2017-03

CONDITIONS: Neuroendocrine Tumors
Keywords: low-grade neuroendocrine tumors; lithium
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Lithium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lithium (Experimental): Lithium carbonate will be dosed on a flat scale of mg/day and not by weight or body surface area (BSA). Lithium carbonate will be provided as a 300mg tablet and will be taken daily without breaks in treatment.
  Interventions: Drug: Lithium Carbonate

INTERVENTIONS:
Drug: Lithium Carbonate — Lithium 300mg PO TID escalating to a lithium level of 0.8-1.2. Lithium carbonate will be administered the first week at 300 mg flat dose three times each day. A serum lithium level will be checked after 4-5 days of treatment by drawing a blood sample prior to the morning dose of lithium. Evaluate every 8 weeks.

SUMMARY:
The purpose of this study is to learn more about the effectiveness and side effects of lithium treatment for subjects with low-grade neuroendocrine tumors.

DETAILED DESCRIPTION:
Lithium 300mg by mouth, three times daily, escalating to a lithium level of 0.8-1.0; Continue until progressive disease/unacceptable toxicity;Evaluate q 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically confirmed metastatic low-grade neuroendocrine neoplasms. Small cell lung cancers, paragangliomas and pheochromocytomas are excluded. Pathologic diagnosis must be confirmed at the University of Wisconsin Carbone Cancer Center (UWCCC). Grading must be confirmed by pathologic review performed at UWCCC.
* Must have measurable disease
* Must have radiographic evidence of disease progression following any prior systemic therapy, chemoembolization, bland embolization, surgery, or observation.
* Must be ≥ 4 weeks from the completion of major surgery, chemotherapy, or other systemic therapy or local liver therapy to study registration
* Must be ≥ 3 weeks from the completion of radiation therapy to study registration
* The following laboratory values are to be obtained within 14 days prior to registration: Absolute neutrophils count (ANC) ≥ 1000/mm3; Platelets ≥ 75,000/mm3; Hemoglobin ≥ 8.0 g/dL; Total bilirubin less than or equal 2.0 X the upper limit of normal (ULN); AST less than or equal to 3 X ULN or less than or equal 5 X ULN if liver metastases are present; Creatinine less than or equal ULN; Serum sodium within normal limits
* PS = 0-2
* Capable of understanding the investigational nature, potential risks and benefits fo the study and able to provide valid informed consent.
* Must have available tissue specimens to be analyzed for pathologic confirmation.
* Age ≥ 18 years.
* Women must not be pregnant or lactating.
* Women of childbearing potential and sexually active males are required to use an accepted and effective method of contraception.
* Patients must not have known history of allergic reactions or adverse reactions to Lithium or derivatives.
* Patients are not allowed to be on concurrent chemotherapy or radiation therapy.
* Patients are excluded if they have any of the following:

Gastrointestinal tract disease resulting in an inability to take oral medication (i.e. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, bowel obstruction, or inability to swallow the tablets.

History of hypothyroid disease Significant, active cardiac disease

* Patients must not be taking the following medications: diuretics, ACE inhibitors, NSAIDs (except aspirin or sulindac), neuroleptics, tetracycline, COX2 (cyclooxygenase-2) inhibitors, citalopram, clovoxamine, escitalopram, femoxetine, fluoxetine, fluvoxamine, paroxatine, sertraline, and zimeldine.
* Must be willing to undergo a tumor biopsy pre and post therapy.
* Patients with a concurrent malignancy are allowed on study as long as the patient is not undergoing active treatment for their disease.
* Patients already taking Lithium for any reason are not allowed on study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noelle LoConte, MD, Principal Investigator — University of Wisconsin, Madison; Herbert Chen, MD, Study Chair — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- [Result] Lubner SJ, Kunnimalaiyaan M, Holen KD, Ning L, Ndiaye M, Loconte NK, Mulkerin DL, Schelman WR, Chen H. A preclinical and clinical study of lithium in low-grade neuroendocrine tumors. Oncologist. 2011;16(4):452-7. doi: 10.1634/theoncologist.2010-0323. Epub 2011 Mar 10. PMID 21393344
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled participants with low grade neuroendocrine tumors (NETs) from July 2007 through May 2009.
Groups:
- Lithium: Lithium carbonate was dosed on a flat scale of mg/day and not by weight or body surface area (BSA). Lithium carbonate was provided as a 300mg tablet and was taken daily without breaks in treatment.
  Lithium Carbonate: Lithium 300mg PO TID escalating to a lithium level of 0.8-1.2. Lithium carbonate was administered the first week at 300 mg flat dose three times each day. A serum lithium level was checked after 4-5 days of treatment by drawing a blood sample prior to the morning dose of lithium. Evaluated every 8 weeks.
Period: Overall Study
Arm/Group | Lithium
Started | 15
Completed | 10
Not Completed | 5
Not completed — Death | 5

BASELINE CHARACTERISTICS:
Population: Participants with histologically confirmed metastatic low-grade neuroendocrine neoplasms were enrolled.
Arm/Group | Lithium
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate Measured by the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR) >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >=20% increase in the sum of the longest diameter of target lesions; Stable Disease (SD), small changes that do not meet the above criteria.
Time Frame: Up to 4 years
Measure: Number; unit: participants
Arm/Group | Lithium
Number analyzed (Participants) | 15
participants
  Complete Response (CR) | 0
  Partial Response (PR) | 0
  Progressive Disease (PD) | 0
  Stable Disease (SD) | 8

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Progression free survival is measured from the date of entry on the study to the appearance of new metastatic lesions or objective tumor progression. If a participant did not experience an event of disease progression or death at the time of analysis (03/10/2011), then the patient's data was censored at the date of the last available evaluation.
Time Frame: Up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lithium
Number analyzed (Participants) | 15
months | 4.50 [2.99 to 4.50]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival for a participant is defined as the number of days from the day of first Lithium administration to the participant's death. As of the time of analysis (03/10/2011), median overall survival duration was not reached.
Time Frame: Up to 4 years
Population: The median OS time had not been reached.
Measure: Median (Full Range); unit: participants
Arm/Group | Lithium
Number analyzed (Participants) | 15
participants | NA [NA to NA] — 50% of participants had not died at the time that the final statistics were run.

ADVERSE EVENTS:
Time Frame: Adverse event data were collected on or after Day 0 through 4 years.
Description: Adverse events were reported in a routine manner at scheduled times during the trial. Additionally, certain adverse events were reported in an expedited manner for more timely monitoring of patient safety and care.
Arm/Group | Lithium
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium (N=15)
Creatinine (Investigations) | 1 (1)
Glucose (Metabolism and nutrition disorders) | 1 (1)
Hemoglobin (Investigations) | 1 (1)
Ileus, GI (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 2 (3)
Sodium (Investigations) | 1 (1)
Stricture/stenosis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium (N=15)
Abdominal pain (Gastrointestinal disorders) | 9 (14)
Acute cholecystitis (Hepatobiliary disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (5)
Anorexia (Gastrointestinal disorders) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cognitive disturbance/confusion (Psychiatric disorders) | 2 (2)
Cold (General disorders) | 1 (1)
Cold sensation in hands (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine (Investigations) | 4 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 7 (15)
Dizziness (Nervous system disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema (General disorders) | 1 (1)
Elevated TSH (Endocrine disorders) | 1 (2)
Elevated white blood count (Blood and lymphatic system disorders) | 1 (1)
Emotional changes (General disorders) | 1 (1)
Fatigue (General disorders) | 11 (20)
Fever (General disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Frequency (Renal and urinary disorders) | 1 (1)
Gas pain (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
High ALT (Investigations) | 1 (1)
High AST (Investigations) | 1 (1)
High INR (Investigations) | 1 (1)
High Parathyroid Hormone (Endocrine disorders) | 1 (2)
Hot flashes (Vascular disorders) | 1 (1)
Hyperbilirubinemia (Investigations) | 1 (8)
Hypercalcemia (Investigations) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (15)
Hyperthyroidism (Endocrine disorders) | 1 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (5)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Increased gas (Gastrointestinal disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (4)
Ischemia of small bowel leading to necrosis (Vascular disorders) | 1 (1)
Low Anion Gap (Metabolism and nutrition disorders) | 1 (2)
Low EGFR (Renal and urinary disorders) | 1 (1)
Lymphopenia (Investigations) | 4 (9)
Memory Impairment (Nervous system disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (9)
Panic Attacks (General disorders) | 1 (1)
Puritis (Skin and subcutaneous tissue disorders) | 1 (1)
Shaky legs (Musculoskeletal and connective tissue disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stricture of mesenteric artery (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (9)
Tremors (Nervous system disorders) | 5 (6)
Unsteady Gait (Musculoskeletal and connective tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No